CLINICAL TRIAL: NCT03595111
Title: Does Intraoperative Myocardial Biopsy Have Any Prognostic Value in Predicting Myocardial Protection After Congenital Cardiac Surgery
Brief Title: Myocardial Biopsy in Congenital Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate Profossor of Anesthesiology, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB00008715964
Record Dates: First submitted 2018-07-12; First posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Myocardial Protection
Keywords: Cardiac Protection; Pediatric; Myocardial biopsy; Cardiopulmonary Bypass

STUDY DESIGN:
Intervention Model Description: Myocardial cell edema either focal or diffuse was detected in histopathological examination in pediatric patients undergoing total repair of Tetrology of Fallout
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Myocardial biopsy (Experimental): The specimens were classified into three categories: normal, focal hydropic change and diffuse hydropic change.
  Interventions: Procedure: myocardial biopsy

INTERVENTIONS:
Procedure: myocardial biopsy — Myocardial cell edema either focal or diffuse was detected in histopathological examination

SUMMARY:
Despite major advances in the technical aspects of surgical repair of congenital heart diseases, perioperative myocardial damage with low cardiac output remains the most common cause of morbidity and death after repair of congenital heart lesions.

DETAILED DESCRIPTION:
Myocardial sample was obtained from the endocardial surface of the right ventricle and placed in formalin until examination under light microscopy for detection of myocyte cellular edema as a marker of ischemic changes.

ELIGIBILITY:
Inclusion Criteria:

Scheduled cardiac surgery requiring cardioplegic arrest with expected cross clamp time>45 minutes.

Hemodynamic stability.

Exclusion Criteria:

Previous cardiac surgery. Urgent or emergent cases. Any known allergies to components of either cardioplegia solutions.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Myocardial biopsy | within 24 hours
  Myocardial cell edema either focal or diffuse was detected in histopathological examination

SECONDARY OUTCOMES:
The inotropic score | within one month
  1 point is assigned for each mcg/kg/min of dopamine and dobutamine, and 10 points is assigned for each 0.1 mcg/kg/min of epinephrine, norepinephrine, and phenylephrine. (i.e. 1 point is assigned for each 10 ng/kg/min of epinephrine, norepinephrine, and phenylephrine.
Serum cardiac troponin level | first 24 hours
  Samples for troponin I levels at baseline, 6, 12 and 24 hours after aortic cross-clamping.
30-day mortality | 30 days
  number of patients died
Type of cardiac rhythm on return | within 24 hours
  Type of cardiac rhythm on return

IPD SHARING:
Plan to Share IPD: No